CLINICAL TRIAL: NCT04974892
Title: Investigating the Role of Neutrophils in Aspirin Treatment for Women at High Risk of Preeclampsia
Brief Title: Aspirin and Neutrophils in Preeclampsia
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 294761
Record Dates: First submitted 2021-05-21; First posted 2021-07-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia; Neutrophil; Immunology; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low dose aspirin: high-risk women given LDA at ≤16 weeks.
  Interventions: Diagnostic Test: Blood test
- Non responders to low dose aspirin: high-risk women who have not responded to LDA and have gone on to develop PE.
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Blood tests will be taken at 12, 20, 28 and 36 weeks gestation to assess the immune profile and omic profile.

SUMMARY:
The exact mechanisms by which aspirin prevents the development of preeclampsia in high-risk patients are currently not fully known. Furthermore, a small proportion of high-risk patients who are on low-dose aspirin (LDA) still go on to develop preeclampsia (PE).

This longitudinal observational study will assess the immune profile in participants who are taking low dose aspirin (LDA) in pregnancy. As part of routine care, patients at high risk of developing preeclampsia are treated with LDA from 16 weeks gestation.

The study will be conducted at Barts Health National Health Service (NHS) Trust. The study population will comprise of 2 groups of participants:

1. Those who respond to LDA and do not develop preeclampsia (responders)
2. Participants who do not respond to LDA and develop preeclampsia (non responders)

Participants will be consented at their booking appointment. Participants will be eligible if they have a singleton pregnancy and are aged over 18 years. They will have an additional blood sample taken at 12, 20, 28 and 36 weeks gestation.

The blood samples will be tested to assess immune cell function, metabolism and genetics. This will identify cumulative changes in immunobiology at key time points in pregnancy.

DETAILED DESCRIPTION:
The exact mechanisms by which aspirin prevents the development of PE in high-risk patients are currently not fully known. Furthermore, a small proportion of high-risk patients who are on low-dose aspirin still go on to develop PE. This is a big unmet need because although it is known that this treatment is working for some patients, it is not known how it's working in these patients and also why a proportion of patients don't respond to this treatment. If the key mechanisms by which aspirin treatment is beneficial in patients at high risk of PE can be identifies, this will lead to better information for clinicians of why this treatment works and this could then be conveyed to the patient. Moreover, if key differences can be identified between aspirin responders and non-responders, novel therapeutic targets could be developed that could work for all patients at high risk of PE.

One of the main anti-inflammatory actions of aspirin is the release of aspirin-triggered lipoxin (ATL). The receptor for ATL (FPR2/ALX) is highly expressed on neutrophils, suggesting that the anti-inflammatory action of this drug is mediated via neutrophils. The investigators have previously shown that neutrophils are important in mediating anti-inflammatory responses in PE. Thus, taken together, the hypothesis is that neutrophils are key to understanding the mechanisms involved in the use of low-dose aspirin (LDA) treatment in patients at high risk of developing PE and key to understanding why this treatment does not work in some high-risk patients. This hypothesis will be addressed by two objectives both of which will entail in-depth profiling of neutrophils.

ELIGIBILITY:
Inclusion criteria

* Age 18-60 years
* Singleton pregnancy
* Live fetus at 11-13 weeks of gestation
* Informed, written consent
* Upper age of 60 years
* Patient taking low dose aspirin as standard of care

Exclusion criteria

* Unwilling or unable to give consent
* Participants who are unable to understand written English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high risk of developing preeclampsia in pregnancy who are started on low dose aspirin at ≤16 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To longitudinally define the neutrophil profile in high-risk patients given low dose aspirin (LDA) at ≤16 weeks. | 2 years
  To address the first objective, to assess the neutrophil profile in high-risk patients given LDA at ≤16 weeks, a longitudinal analyses will be undertaken of neutrophils taken from participants at high-risk of PE (as identified at their pregnancy booking appointment). The first blood test will occur prior to aspirin commencement and be repeated at 3 other time points in pregnancy. These longitudinal analyses will identify cumulative changes in neutrophils following the commencement of aspirin treatment and pinpoint key timepoints of aspirin on neutrophil biology.
To define the neutrophil profile in a cohort of high-risk patients who have not responded to low dose aspirin (LDA) and have gone on to develop PE. | 2 years
  To address the second objective (to assess the neutrophil profile in a cohort of high-risk patients who have not responded to LDA and have gone on to develop PE), 20 LDA non-responders subsequently develop PE will be identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No